CLINICAL TRIAL: NCT04095689
Title: Phase II Study of Docetaxel Chemotherapy With Pembrolizumab and Interleukin-12 Gene Therapy in Patients With Anthracycline- Refractory Triple Negative Breast Cancer (INTEGRAL)
Brief Title: Docetaxel Chemotherapy and Pembrolizumab Plus Interleukin-12 Gene Therapy in Triple Negative Breast Cancer
Acronym: INTEGRAL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopping rules met per protocol, trial will be terminated
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Polly A. Niravath, MD, Professor of Medicine in Oncology, Academic Institute, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00028602
Record Dates: First submitted 2019-09-18; First posted 2019-09-19 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Triple Negative Breast Cancer; Anthracycline-refractory TNBC
Keywords: triple negative breast cancer, neoadjuvant, pembrolizumab; anthracycline-refractory TNBC
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Docetaxel; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): docetaxel chemotherapy and pembrolizumab plus IL-12 gene therapy.
  Interventions: Drug: Docetaxel; Drug: Pembrolizumab; Drug: IL-12 gene therapy

INTERVENTIONS:
Drug: Docetaxel — Microtubule-targeting drug (inhibits microtubule depolymerization)
  Other Names: Taxotere
Drug: Pembrolizumab — Programmed cell death-1 (PD-1) inhibitor
  Other Names: Keytruda
Drug: IL-12 gene therapy — Adenoviral-mediated IL-12

SUMMARY:
The purpose of this research study is to test the safety and effectiveness of docetaxel chemotherapy and pembrolizumab plus adenoviral-mediated interleukin-12 (ADV/IL-12) gene therapy in patients with anthracycline-refractory, triple negative breast cancer (TNBC).

DETAILED DESCRIPTION:
The purpose of this study is to learn how triple negative breast cancer (TNBC) responds to the use of chemotherapy, pembrolizumab, and gene therapy together in patients who have previously not responded to treatment. We will also look at the effects, good or bad, the study therapy has on you and your TNBC.

Chemotherapy given before breast cancer surgery is called neoadjuvant chemotherapy. It shrinks the breast tumor, so it is easier to remove during surgery. Docetaxel is often used for the neoadjuvant treatment of breast cancer. Unfortunately, a lot of breast tumors do not shrink with docetaxel chemotherapy treatment. Docetaxel chemotherapy is standard care for TNBC.

Pembrolizumab is a type of treatment that stimulates your own immune system to attack cancer cells. Your immune system is normally your body's first defense against threats like cancer. However, sometimes cancer cells produce signals that prevent the immune system from detecting and killing them. Pembrolizumab helps your immune system so it can detect and attack cancer cells. Chemotherapy plus pembrolizumab has been shown to be better than chemotherapy alone for shrinking breast tumors before surgery.

To help increase the tumor-shrinking activity of docetaxel chemotherapy and pembrolizumab, you will be given more treatments, Interleukin-12 (IL-12) gene therapy This treatments will be used to boost the cancer-fighting ability of your immune system. Thus, the use of IL-12 gene therapy with docetaxel chemotherapy and pembrolizumab may make your immune system work harder to shrink your tumor. IL-12 is a substance that is normally made by certain immune cells in the body. IL-12 stimulates T cells, a special type of immune cell in the blood, to respond to threats to your body like cancer.

After you finish the study treatment, you will have your breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the trial only if all of the following criteria apply:

1. The patient (or legally acceptable representative if applicable) provides written informed consent for the trial.
2. Female ≥ 18 years of age on the day of informed consent signing.
3. Histologically confirmed triple negative breast cancer is defined as estrogen receptor (ER), progesterone receptor (PR), and HER2 negative. ER/PR negativity is defined as <10% IHC staining of any intensity.

HER2 negativity is defined as the following per the 2018 American Society of Clinical Oncology and College of American Pathologists guidelines.

4. Refractory to standard neoadjuvant anthracycline-containing chemotherapy regimen, demonstrated on MRI.

5. Bilateral breast cancers that individually meet eligibility criteria are allowed.

6. Prior immunotherapy treatment allowed. 7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. 8. Adequate organ function as defined in Table 1. All screening labs should be performed within 28 days of trial treatment initiation.

9. Cardiac ejection fraction ≥45%. 10. A female patient is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

1. Not a woman of childbearing potential (WOCBP) OR
2. A WOCBP who agrees to follow the contraceptive guidance in during the treatment period and for at least 120 days after the last dose of trial treatment. WOCBP must have a negative serum pregnancy test (β-human chorionic gonadotropin [β-HCG]) within 72 hours prior to trial treatment administration.

   11. Willing to provide biopsy tissue as required by the trial. 12. Willing and able to comply with the protocol for the duration of the trial including undergoing treatment and scheduled visits and examinations.

   Exclusion Criteria:
   1. History of poorly controlled hypertension (defined as systolic blood pressure >150 mmHg). Patients whose hypertension has been well controlled on the same treatment for 1 year prior to Cycle 1, Day 1 are eligible. Only patients on single-agent antihypertensive therapy are allowed.
   2. History of New York Heart Association class III or greater cardiac disease.
   3. History of myocardial infarction, stroke, ventricular arrhythmia, or greater than first-degree conduction defect within the past 12 months.
   4. History of congenital QT prolongation.
   5. Absolute corrected QT interval of >480 msec in the presence of potassium >4.0 mEq/L and magnesium >1.8 mg/dL.
   6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to trial treatment administration.

   NOTE: Patients who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

   8. Concurrent use of any complementary or alternative medicines. 9. Concurrent use of inhibitors or inducers of cytochrome P450 (CYP)3A4 and CYP2D6 10. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (dose exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to trial treatment administration.

   11. Known history of active tuberculosis (Bacillus Tuberculosis). 12. Known or suspected hypersensitivity to any component or excipient of the proposed regimen (docetaxel chemotherapy, gene vector, pembrolizumab).

   13. Patients must have recovered from all AEs due to previous therapies to ≤ Grade 1 or baseline. Patients with ≤ Grade 2 neuropathy may be eligible. If patient received major surgery, she must have recovered adequately from the toxicity and/or complications from the intervention prior to starting the trial treatment.

   14. Known additional malignancy that is progressing or requires active treatment. NOTE: Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or cervical cancer in situ that have undergone potentially curative therapy are not excluded.

   15. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

   16. History of (noninfectious) pneumonitis that required steroids or current pneumonitis.

   17. Active infection requiring systemic therapy. 18. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.

   19. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

   20. Pregnant or breastfeeding, or expecting to conceive children within the projected duration of the trial, starting with the prescreening or screening visit through 120 days after the last dose of trial treatment.

   21. Known history of human immunodeficiency virus (HIV). 22. Known history of hepatitis B (defined as hepatitis B surface antigen reactive) or known active hepatitis C virus (HCV; defined as HCV RNA [qualitative] is detected) infection.

   23. Received a live vaccine within 30 days prior to trial treatment administration. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was consented on 5/12/2021 and the last patient was consented on 5/16/2023. The final patient was off study on 5/3/2024.
Period: Overall Study
Arm/Group | Experimental
Started | 8
Completed | 3
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 56 [32 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response (pCR) Rate of Docetaxel Chemotherapy and Pembrolizumab Plus IL-12 Gene Therapy
Description: To determine the pCR rate of docetaxel chemotherapy and pembrolizumab plus IL-12 gene therapy in patients with TNBC per RECIST v1.1 assessed by CT Scan or MRI. CR: Disappearance of all target lesions. PR: at least a 30% decrease in the sum of the longest diameter of target lesions, using the baseline sum longest diameter as a reference. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, using the smallest sum longest diameter as a reference. PD: At least a greater than or equal to 20% increase in the sum of the longest dimensions of the target lesions taking as a reference the smallest sum of the longest dimensions recorded since the treatment started, or the appearance of one or more new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Clinical PD: Patients who in the opinion of the treating PI have clinical evidence of PD may be classified as having PD
Time Frame: 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 8
Participants | 1

2. Secondary Outcome: Number of Participants With Treatment-related Adverse Events
Description: To determine the number of participants with treatment-related adverse events, as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events v5.0
Time Frame: 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 8
Participants | 8

ADVERSE EVENTS:
Time Frame: At the time of informed consent through 90 days after last treatment dose, approximately 26 weeks (28 Days through screening + 4 - 21 day cycles + 90 days after last treatment dose on cycle 4 day 1)
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 2/8
Serious Adverse Events (participants affected / at risk) | 6/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=8)
Ferbile Neutropenia (Blood and lymphatic system disorders) | 3 (3) — Definitely Related to Treatment
Hepatic Biliary disorders, other (Hepatic Toxicity) (Hepatobiliary disorders) | 1 (1) — Possibly Related to Treatment
Sepsis (Infections and infestations) | 2 (2) — Related to Treatment
Fatigue (General disorders) | 1 (1) — Definitely Related to Treatment
Aspartate aminotransferase increased (Transaminitis) (Investigations) | 1 (1) — Possibly Related to Treatment
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Possibly Related to Treatment
Thromboembolism (Vascular disorders) | 1 (1) — Not Related to Treatment
Right Breast Hematoma (Vascular disorders) | 1 (1) — Not Related to Treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=8)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) — Not Related to Treatment
Alanine aminotransferase increased (Investigations) | 2 (2) — Possibly Related to Treatment
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly Related to Treatment
Aspartate aminotransferase increased (Investigations) | 2 (2) — Possibly Related to Treatment
Headache (Nervous system disorders) | 2 (2) — Related to Treatment
Bone Pain (Musculoskeletal and connective tissue disorders) | 3 (3) — 1 event was related, 2 events were not related
Chills (General disorders) | 3 (3) — Related to Treatment
Constipation (Gastrointestinal disorders) | 3 (3) — Related to Treatment
Diarrhea (Gastrointestinal disorders) | 3 (3) — Possibly Related to Treatment
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Not Related to Treatment
Edema Limbs (General disorders) | 2 (3) — Unlikely Related to Treatment
Fatigue (General disorders) | 5 (5) — Possibly Related to Treatment
Fever (General disorders) | 5 (5) — Related to Treatment
Nail Discoloration (Skin and subcutaneous tissue disorders) | 1 (1) — Related to Treatment
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) — Possibly Related to Treatment
Hypotension (Vascular disorders) | 1 (1) — Not Related to Treatment
Breast Infection (Left) (Infections and infestations) | 1 (1) — Not Related to Treatment
Dysgeusia (Nervous system disorders) | 1 (1) — Possibly Related to Treatment
Mucositis oral (Gastrointestinal disorders) | 3 (3) — Possibly Related to Treatment
Nausea (Gastrointestinal disorders) | 1 (1) — Possibly Related to Treatment
Peripheral Sensory Neuropathy (Nervous system disorders) | 3 (6) — Related to Treatment
Ocular Migraine (Nervous system disorders) | 1 (1) — Not Related to Treatment
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) — Possibly Related to Treatment
Right Axillary Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Unlikely Related to Treatment
Right Leg Discoloration (Skin and subcutaneous tissue disorders) | 1 (1) — Not Related to Treatment
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) — Possibly Related to Treatment
Skin Infection (Infections and infestations) | 1 (1) — Not Related to Treatment
Tachycardia (Cardiac disorders) | 2 (3) — 1 Related to Treatment, 2 Not Related to Treatment
Upper Respiratory Infection (Infections and infestations) | 1 (1) — Not Related to Treatment
Urinary tract infection (Infections and infestations) | 1 (1) — Not Related to Treatment
Vomiting (Gastrointestinal disorders) | 1 (1) — Not Related to Treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT04095689/Prot_SAP_000.pdf